CLINICAL TRIAL: NCT00707213
Title: FDG-PET/CT In the Evaluation of Persistent Febrile Neutropenia in Cancer Patients
Brief Title: FDG-Positron Emission Tomography (PET)/CT In the Evaluation of Persistent Febrile Neutropenia in Cancer Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding from the NIH ended and not all patients had been accrued
Sponsor: University of Utah (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HCI22418; R21CA128228-01 (NIH)
Record Dates: First submitted 2008-06-25; First posted 2008-06-30 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Participants (Experimental): All Participants will be assessed by FDG-PET to identify possible sites of infection
  Interventions: Drug: [18F]fluoro-2-deoxy-D-glucose (FDG)

INTERVENTIONS:
Drug: [18F]fluoro-2-deoxy-D-glucose (FDG) — FDG-PET/CT scan-The scans that will be done with a radioactive sugar ([18F]fluoro-2-deoxy-D-glucose) and positron emission tomography (FDG-PET/CT). These scans will help to identify areas of possible infection.
  Other Names: FDG; [18F]FDG; FDG-PET/CT

SUMMARY:
Patients must be currently treated at the Huntsman Cancer Institute or Intermountain Primary Children's Medical Center to be eligible for this study.

Although there have been many advances in the assessment and treatment of infections responsible for febrile neutropenia in cancer patients, it still remains a common complication of cancer therapy and accounts for the majority of chemotherapy-associated deaths. This National Cancer Institute (NCI) funded proposal using the R-21 Quick-Trials Exploratory Grant mechanism is to conduct an exploratory/pilot project in a group of patients with persistent febrile neutropenia to provide critical information that will support the concept, and aid in the design, of a larger multi-center clinical trial. The ultimate goal of our interdisciplinary team of oncologists, infectious diseases experts, imagers, and biostatisticians is to conduct a prospective, multi-center trial to establish the utility and cost-effectiveness of PET/CT using the widely available glucose analogue [18F]fluoro-2-deoxy-D-glucose (FDG) in identifying sites of infection in cancer patients with persistent febrile neutropenia without an obvious identifiable source thus improving targeted therapy.

DETAILED DESCRIPTION:
What is the significance of this project? The significance is two fold: (1) the serious nature of the clinical condition that it addresses, and (2) in the potential ease and safety by which this approach could be translated to clinical practice. Although there have been many advances in treatment modalities related to febrile neutropenia, it still remains a common complication of cancer therapy and accounts for the majority of chemotherapy-associated deaths (Sipsas 2005). The broad-spectrum therapeutic management of febrile neutropenia is often "shotgun" in its approach, without a clear source to allow target-specific therapy. The subpopulation of patients with febrile neutropenia that present the greatest problem is that with persistent febrile neutropenia > 5 days despite broad spectrum antibiotics, and without an identifiable source of infection. As noted previously, however, the definition of persistence is changing in medical practice. Currently medical professionals are ordering diagnostic imaging studies such as CT scans earlier due to the need to localize a site of infection and use the most appropriate antibiotic therapy. Without a target, multi-drug antibiotic therapy in these patients can continue for many weeks. The drugs are often toxic, with substantial side effects. Hospitalization is extended. The cost of broad spectrum hospital course of antibacterial and antifungal drugs is in the range of multiples of $10,000, and the cost of extended hospitalization to treat an unknown infection in a patient with persistent febrile neutropenia may be multiples of $100,000. Chemotherapy may be suspended or discontinued, with risk of development of chemo-resistant tumor cells. Conventional imaging methods are limited in evaluation of febrile neutropenia due to lack of anatomic changes. The lack of sufficient white cells to mount an inflammatory reaction compromises detection of sites of infection by radiography or CT.

Because white cell number is severely reduced, the use of labeled white cell scans is often precluded. If FDG-PET/CT can provide a likely anatomic site for targeted antibiotic therapy in this specific high risk population, it is possible that morbidity/mortality from infection and antibiotic side effects may be minimized, hospitalization days may be reduced, and effective anti-cancer therapy may be continued without interruption. Although FDG-PET/CT is not cheap, the ultimate result may be highly cost-effective.

Our oncologist and infectious diseases co-investigators predict that a tissue diagnosis can be obtained in at least 80% of all FDG-PET/CT or CT findings that are suspicious for infection in children and 50% in adults. This confirmatory tissue diagnosis will serve as the "gold standard" to assess the effectiveness of FDG-PET/CT in finding a source of infection.

Additional confirmatory factors will include clinical response to targeted therapy and resolution of associated radiographic or CT findings. The data will be evaluated to address the following questions, which are the sub-aims of the funded proposal:

1. How effective is FDG-PET/CT in identifying sites of infection in patients with febrile neutropenia without an obvious cause?
2. To what degree does FDG-PET/CT improve detection of sites of infection over CT alone?
3. What FDG-PET/CT imaging variables best predict the presence of infection at a specific site (e.g. standardized uptake value (SUV), concomitant abnormality on CT)?
4. Can the magnitude of uptake of FDG measured by an SUV at sites of infection predict the identity of the infective agent (bacterial vs. fungal vs. viral)?
5. Does magnitude of uptake at sites of infection correlate with absolute neutrophil count (ANC)?
6. Can a clinical scoring system be developed to identify a population of patients in whom FDG-PET/CT is likely to be most efficacious in identifying sites of infection?

This pilot data will be used to determine whether there is sufficient support for, and to aid in the design of, a large, prospective, multi-center clinical trial to establish the cost-effectiveness and efficacy of FDG-PET/CT in evaluation of febrile neutropenia, compared to patients who are managed by conventional methods.

ELIGIBILITY:
Pediatric patients:

All pediatric subjects will be recruited from Intermountain Primary Children's Medical Center (PCMC). At any point in time, there are 6-10 inpatients at PCMC who are being treated as in-patients for febrile neutropenia. Each day, 2-3 new patients with febrile neutropenia are admitted or transferred to PCMC from hospitals and clinics across the intermountain area. Approximately 3-5 patients per week will be eligible for inclusion in this study (having high-risk persistent febrile neutropenia without an obvious cause). The target for this study is to recruit a minimum of 1-2 pediatric patients per month to the protocol. Therefore, the eligible pediatric patient population should be more than sufficient to meet this goal. Most of these patients are >10 years of age. The vast majority are adolescents and teenagers, because pediatric patients at highest risk for febrile neutropenia are those on high dose methotrexate for high risk leukemia and lymphomas that target adolescents and teenagers. Leukemics constitute the largest percentage of these patients. To be eligible for inclusion, subjects must be admitted for treatment as in-patients for febrile neutropenia, with an absolute neutrophil count (ANC) < 500 cells/mm3, in whom a fever persists without obvious source despite 5 days of broad spectrum antibiotics. Typically, pediatric patients in this category will have been treated with IV Fortaz (ceftazidime). We will also study patients that do not meet the older definition of persistent (> 5 days) fever who for medical reasons an advanced imaging study (typically CT scans) is now medically indicated for localization of a possible site of infection. These patients will have a fever and be neutropenic, however they may not have been febrile for > 5 days. Medical imaging is indicated sooner than the typical 5 days due to the patients condition and need to localize a site of infection.

Exclusion criteria will include inability to undergo a FDG-PET/CT scan without conscious sedation, medical instability that would preclude safe transport to the PET center in the Huntsman Cancer Hospital (PCMC does not have a PET scanner), and a fasting serum glucose > 200 mg/dl. A negative pregnancy test will be required in post-menarche females prior to inclusion.

Adult patients:

All adult subjects will be recruited from the Huntsman Cancer Hospital, patients will be recruited from the general oncology service. As for the pediatric patients, those considered eligible will include those with a documented fever > 5 days despite IV antibiotics, an ANC < 500 cells/mm3, and in patient treatment as a high risk patient. We will also study patients that do not meet the older definition of persistent (> 5 days) fever who for medical reasons an advanced imaging study (typically CT scans) is now medically indicated for localization of a possible site of infection. These patients will have a fever and be neutropenic, however they may not have been febrile for > 5 days. Medical imaging is indicated sooner than the typical 5 days due to the patients condition and need to localize a site of infection. On average, 5-6 patients per week are admitted to the Huntsman Cancer Hospital with the diagnosis of high risk persistent febrile neutropenia. At any one time, there are typically 3-4 adult in patients on the ward with the diagnosis of persistent febrile neutropenia. Of these, approximately 2-3 patients per week will be eligible for inclusion in this study (having persistent febrile neutropenia without an obvious cause). The target for this study is to recruit a minimum of 1-2 adult patients per month to the protocol. Therefore, the eligible adult patient population should be more than sufficient to meet this goal. As with the pediatric population, the majority of these patients have leukemia and lymphoma (50:50). Adult patients may also have multiple myeloma. In these patients, the typical duration of neutropenia is 3-4 weeks. Typically, the initial workup of the adult patients with febrile neutropenia is a chest X-ray, complete blood count (CBC), urinalysis, peripheral and central line blood culture, and additional studies only as directed by symptoms. Initial in-patient treatment for high risk patients is typically with IV meropenem and ceftazidime. If fever persists beyond 5 days without specific localizing signs or symptoms, antibacterials may be changed or added, and antifungals are started (typically amphotericin B or caspofungin), typically persisting until the white count returns to 1000 cell/mm3. Additional imaging studies are not done on a consistent basis for the adults with persistent high-risk febrile neutropenia. Extended imaging is typically done only as symptoms dictate. Typically, a source of infection is found in only 40-50% of patients with febrile neutropenia at our institutions as well as from the literature (Chaimberlain 2005; Hughes 2002; Roguin 1996). In the persistent febrile neutropenia patient despite further and more comprehensive evaluation and assessment a source is identified in only about an additional 10% of these patients.

As with pediatric patients, adult exclusion criteria will include inability to undergo a FDG-PET/CT without conscious sedation, medical instability, a fasting serum glucose > 200 mg/dl, and pregnancy. A negative pregnancy test will be required of all females of reproductive potential prior to inclusion.

Of note, patients from the bone marrow transplant unit will be eligible to participate in this pilot study,. Many of these patients are placed on prophylactic antifungal agents at the time of presentation of neutropenia and fever. This may cause a drug-induced fever in a certain percentage of recipients. For this reason, the clinical picture is clouded however the patients may still have an occult infection. Bone marrow transplant patients will be included in the study as this is an exploratory study and the information gained from assessing the ability of FDG-PET/CT to localize sites of infection in neutropenic, febrile bone marrow transplant patients will be valuable.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-08-21 (Actual); Primary Completion 2010-08-11 (Actual); Study Completion 2010-08-11 (Actual)

PRIMARY OUTCOMES:
The primary goal of this study is to perform FDG-PET/CT scans in approximately 100 cancer patients (both adults and children) with persistent febrile neutropenia where the source of infection has not been identified. | December 2011

CONTACTS AND LOCATIONS:
Overall Officials: John M Hoffman, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States